CLINICAL TRIAL: NCT03149614
Title: Clinical Effects in Cervical Spinal Mobilization Versus Resonant Oscillation Mobilization (POLD) in Neck Pain. A Randomized Clinical Trial.
Brief Title: Clinical Effects in Cervical Spinal Mobilization and Oscillation Mobilization in Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Jaime Salom Moreno, PT, PhD, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: URJC201701
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Manual Therapy; Neck Pain
Keywords: mobilization; resonant oscillation
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spine Mobilizations (Active Comparator): Patients receive spinal mobilizations in grades II to III of central posterior-anterior from cervical and thoracic spine as described Maitland in 2000.
  Interventions: Other: Spine Mobilizations
- Vertebral Resonant Oscillation (POLD method) (Experimental): The vertebral resonant oscillation using the POLD method is similar to spine mobilizations, but there are some differens; the oscillatory movement has a sinusoidal waveform, the frequency used between 1.2 and 2 Hz and the amplitude is similar to "neutral zone" to described by Panjabi 1992.
  Interventions: Other: Vertebral Resonant Oscillation

INTERVENTIONS:
Other: Spine Mobilizations — Patients receive spinal mobilizations in grades II to III of central posterior-anterior from cervical and thoracic spine as described Maitland in 2000
  Arms: Spine Mobilizations
Other: Vertebral Resonant Oscillation — The vertebral resonant oscillation using the POLD method is similar to spine mobilizations, but there are some differens ; the oscillatory movement has a sinusoidal waveform, the frequency used between 1.2 and 2 Hz and the amplitude is similar to "neutral zone" to described by Panjabi 1992.
  Arms: Vertebral Resonant Oscillation (POLD method)

SUMMARY:
The aim of this study is to compare the clinical effects of spinal mobilization versus vertebral resonant oscillation (POLD) in patients with bilateral mechanical neck pain on pain sensitivity and neck pain intensity.

DETAILED DESCRIPTION:
The clinical practice guidelines for manual therapy management the neck pain including the spine mobilization.

The vertebral resonant oscillation using the POLD method is similar to spine mobilizations, but there are some differens; the oscillatory movement has a sinusoidal waveform, the frequency used between 1.2 and 2 Hz and the amplitude is similar to "neutral zone" to described by Panjabi 1992.

The spinal mobilizations has a posterior-anterior vertebral movement for spinous process, described by Maitland 2000.

ELIGIBILITY:
Inclusion Criteria:

* neck pain symptoms of mechanical nature
* age from 18 to 60 years
* bilateral symptoms
* symptoms for at least 3 month of duration

Exclusion Criteria:

* whiplash injury
* previous spine surgery
* diagnosis of cervical radiculopathy or myelopathy
* having undergone any physical therapy intervention in the previous 6 month
* pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-10-25 (Actual)

PRIMARY OUTCOMES:
Changes in pain intensity before and after the intervention | Baseline, one week after the last session, 1 months and 3 months after the last session.
  A 10-point Numerical Pain Rating Scale (NPRS; 0: no pain, 10: maximum pain) will be used to assess the patients' current level of neck pain

SECONDARY OUTCOMES:
Changes in disability before and after the intervention | Baseline, one week after the last session, 1 months and 3 months after the last session.
  Neck Pain Disability Index (NDI)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Rey Juan Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No